CLINICAL TRIAL: NCT01447303
Title: Functional and Quality of Life Outcomes Following Hyaluronic Acid (HA) Viscosupplementation for Knee Osteoarthritis
Brief Title: Functional and Quality of Life Outcomes Following Viscosupplementation for Knee Osteoarthritis
Status: Terminated | Type: Observational
Why Stopped: Inability to recruit subjects
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 293-2009
Record Dates: First submitted 2011-09-29; First posted 2011-10-06 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2014-01

CONDITIONS: Knee Osteoarthritis
Keywords: knee; osteoarthritis; hyaluronic acid; viscosupplementation
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Outcomes following viscosupplemantation: Patients with documented knee osteoarthritis receiving viscosupplementation of the knee.
  Interventions: Other: Subject outcomes following viscosupplementation of the knee

INTERVENTIONS:
Other: Subject outcomes following viscosupplementation of the knee — The study subject outcomes (WOMAC, VAS, SF-36, Chair rise, Stair climb, Six minute walk and Gait analysis) measured at 1, 3, 6 and 12 months following viscosupplementation of the knee

SUMMARY:
This study will compare changes in outcomes following viscosupplementation for knee osteoarthritis.

DETAILED DESCRIPTION:
The specific aims of this study are to compare the changes in knee pain symptoms, physical function, gait parameters and quality of life in persons with knee OA following a standard viscosupplementation injection series of hyaluronic acid (HA) over a one year period.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age or older
* osteoarthritis degeneration, degenerative joint disease or degeneration
* fully cognizant of study procedures
* willing to carefully participate in all study processes and assessments

Exclusion Criteria:

* less that 21 years of age
* allergic reactivity to hyaluronic acid
* current knee infection, infection around injection site or any skin disease
* pregnancy or lactation
* non-ambulatory

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic knee osteoarthritis.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2009-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Decsribes any change from baseline over a period of 12 months; the study subjects will complete the (WOMAC) Index at baseline, 1, 3, 6 and 12 months following the viscosupplementation of the knee.
  The (WOMAC) Index is a multidimensional, self-administered health status instrument for patients with osteoarthritis of the hip or knee. The index is a disease-specific, purpose built, high performance instrument for evaluative research in osteoarthritis clinical trials.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) documentation of the level of knee pain. The (VAS) will describe the change in the level of knee pain from baseline following viscosupplementation of the knee. | The study subjects will complete the (VAS) at baseline, 1, 3, 6 and 12 months following the viscosupplementation of the knee.
  The (VAS) responses are expressed on a ten centimeter line, with 0 representing no pain and 10 cm representing the worst pain possible. The patient places a mark across the line representing where their perceived pain lies, from no pain to severe pain; measured at rest, standing and rising from a chair.
Medical Outcomes Short Form (SF-36); completed to describe any change in perceived Quality of Life (QOL) from baseline following viscosupplementation of the knee. | The study subjects will complete the (SF-36) at baseline, 1, 3, 6 and 12 mos. following viscosupplementation of the knee.
  The (SF-36) is a validated, internationally recognized standard instrument for assessing perceived (QOL) will be used to assess overall (QOL)
Chair Rise Time; describes any change from baseline in time to rise from a chair following viscosupplementation of the knee | The study subjects will complete the chair rise at baseline, 1, 3,6 and 12 mos. following viscosupplementation of the knee.
  Chair rise time is measured as the time required to move from a sitting position to fully standing. The measure will be repeated three times with the fastest time being recorded.
Stair Climb Time; describes any change in the time from baseline to walk up a flight of 12 steps following viscosupplementation of the knee | The study subjects will complete the stair climb at baseline, 1, 3, 6 and 12 mos. following viscosupplementation of the knee.
  The time to walk up one flight of stairs was measured by having the study subjects walk up one flight of stairs consisting of 12 steps as quickly as possible. This test will be repeated after a 2 to 3 minute rest, and the faster of the two trials will be used for data analysis.
Six Minute Walk Test; describes any change from baseline in leg pain following viscosupplementation of the knee. | The study subjects will complete the six minute walk test at baseline, 1, 3, 6 and 12 mos. following viscosupplementation of the knee.
  The study subjects will walk at a self-selected pace around a pre-measured loop for a period of six minutes. Leg pain symptoms and scores will be collected using the (VAS) scale at one minute intervals. Leg pain location and type will be noted using a leg pain diagram and a subjective list of terms to describe the pain.
Gait Analysis; describes any changes in gait from baseline following viscosupplementation of the knee. | The study subjects will complete the gait analysis at baseline, 1, 3, 6 and 12 mos. following viscosupplementation of the knee.
  The study subjects will walk across a 26 foot long portable walkway. The mat is filled with pressure sensors and the output is fed into a software program. The stride length and frequency, the motion of the center of mass moving over the mat and the foot pressures with the walking steps will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Heather K Vincent, Ph.D., Principal Investigator — University of Florida Department of Orthopaedics and Rehabilitation
Locations (1):
- UF&Shands Orthopaedics and Sports Medicine Institute, Gainesville, Florida, United States